CLINICAL TRIAL: NCT04612192
Title: Light Therapy for Chronic Insomnia in General Practice: a Randomized Double Blind Study
Brief Title: Light Therapy for Chronic Insomnia in General Practice
Acronym: Insolux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7348
Record Dates: First submitted 2019-10-18; First posted 2020-11-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Insomnia Chronic; Sleep Disorder; Circadian Rhythm Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Chronobiology Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active light (Experimental): Active light
  Interventions: Device: Active luminette
- Placebo light (Placebo Comparator): Placebo light
  Interventions: Device: Placebo luminette

INTERVENTIONS:
Device: Active luminette — receive an active light using glasses of 1500 lux (an average of 180 photons/s/cm2, with a maximum wavelenght at 468 nm), 30-minute long light therapy in the morning, in a time period defined by sleep log and chronotype questionnaire, on a 4-week period
  Arms: Active light
Device: Placebo luminette — receive a placebo light using glasses (an average of n photons/s/cm2, single- band spectrum with a narrow peak at 660 nm under 50 lux), with the same modality as the experimental group
  Arms: Placebo light

SUMMARY:
* Sleep disorders, especially insomnia
* Attention deficits (or disorders), daytime somnolence and drug dependence
* The goal is to evaluate whether light therapy could be used as an efficient alternative treatment with direct application in general practice

DETAILED DESCRIPTION:
Insomnia affects 15 to 20% of the general French adult population and increases with age. General practitioners (GPs) are the first confronted to sleep disorders, especially insomnia.

Cognitive-behavioral therapies (CBT) have proven effective, but their implementation in everyday practice is limited, and alternative treatments are still needed.

Light not only has a great influence on the sleep-wake cycle and alertness, but also on mood and cognitive functions.

The administration time of light condition will be calculated for each individual in a modality that has no impact on the circadian phase.

Study will be conduct on an outpatient basis in general practice

ELIGIBILITY:
Inclusion Criteria:

* Complaining of chronic insomnia according to ICSD-3 (International Classification of Sleep Disorders) criteria and/or taking hypnotics at least 3 nights per week for more than 3 months.
* Non-hypnotic medication: stable medication during one month preceding the inclusion and for the 8 weeks of the study.
* Compliance with the treatment: the patient is able to have light therapy during the required time and at the agreed schedule.

Exclusion Criteria:

* Severe psychiatric disorder (severe major depression, schizophrenia, bipolar disorder), obvious acute psychiatric comorbidity.
* Untreated intrinsic sleep pathology: sleep apnea syndrome based on clinical criteria: STOP-BANG questionnaire score, restless legs syndrome manifesting more than 2 times a week and/or requiring treatment.
* Mild to severe dementia.
* Neurodegenerative sleep troubles
* Severe intercurrent pathology.
* Ophthalmic troubles presenting a contraindication to light therapy: retinopathy, age-related macular degeneration, diabetic retinopathy, macular hole, epiretinal membrane); lens opacifications (cataract) justifying surgery (correction of poor visual acuity, visual discomfort); glaucomatous and non-glaucomatous optic neuropathy resulting in visual impairement.
* Toxicomania, chronic alcoholism.
* Secondary insomnia linked to somatic non-stabilized pathology.
* Elements influencing circadian rhythm
* Pregnancy, breastfeeding.
* Participation in another interventional clinical trial which includes an exclusion period
* No information could be given to the patient (subject faces emergency situation, comprehension difficulties, etc.)
* Patient under guardianship
* Non hypnotic treatment potentially inducing a level 3 sleepiness one week before

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — randomisation by sex
Enrollment: 240 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Difference of sleep efficiency between active and placebo light condition | Before light therapy
  ratio of total sleep time on total time in bed in measured with actimetry
Difference of sleep efficiency between active and placebo light condition | After 4 weeks of light therapy
  ratio of total sleep time on total time in bed measured with actimetry

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University of Nantes, Nantes
  - CHU Reims, Reims
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No